CLINICAL TRIAL: NCT06956469
Title: BmemHLA : Origins of the Heterogeneity of the Anti-HLA Memory B Cells in Kidney Transplantation
Acronym: BmemHLA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2023/39
Record Dates: First submitted 2025-04-25; First posted 2025-05-04 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Kidney Transplantation; Immunology
Keywords: Kidney; Memory B Cell; Anti-HLA antibodies; Allogeneic events; Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Sensitizing events : Pregnancy (Active Comparator): Patients who have been pregnant
  Interventions: Other: Identification of types of anti-HLA-specific memory LBs
- Sensitizing events : Previous transplantation with thrombosis (Active Comparator): Previous transplantation with early transplantectomy due to thrombosis
  Interventions: Other: Identification of types of anti-HLA-specific memory LBs
- Sensitizing events : Previous transplantation with antobody (Active Comparator): Previous transplantation with antibody-mediated rejection
  Interventions: Other: Identification of types of anti-HLA-specific memory LBs
- Whitout any sensitizing event (Active Comparator): Patients who have anti-HLA antibodies without any sensitizing event identified
  Interventions: Other: Identification of types of anti-HLA-specific memory LBs
- Sensitizing events : Transfusion (Active Comparator): Patients who received a blood transfusion
  Interventions: Other: Identification of types of anti-HLA-specific memory LBs

INTERVENTIONS:
Other: Identification of types of anti-HLA-specific memory LBs — Using blood sample, it will be perform single cell RNA sequencing of sorted anti-HLA B cells, identified with HLA tetramers, of five groups of patients based on their immunization histories. It will be further perform a phenotypic characterization of the tetramer+ anti-HLA B cells using spectral cytometry to study their nature and identify novel markers of memory subgroups.

SUMMARY:
This study will describe the transcriptomic and phenotypic characteristics of anti-HLA memory B cells by comparing five groups of patients awaiting renal transplantation: patients with a single history of pregnancy, transfusion or failure of a first renal transplant requiring transplantectomy within 3 months of transplantation, or after 3 months, and patients without an immunizing allogeneic event. The hypothesis is that these five contexts induce different types of memory B cells with different modalities of reactivation and post-transplant pathogenicity.

DETAILED DESCRIPTION:
In kidney transplantation, the production of anti-HLA antibodies directed against the donor (DSA for Donor Specific Antibodies) can be responsible for humoral rejection, the main cause of long-term graft loss. Reactivation of anti-HLA memory B cells after transplantation is thought to play a major role in DSA production and the occurrence of humoral rejection. The investigators hypothesize that the nature and the function of anti-HLA memory B cells could differ depending on how they were initially generated. Several sensitizing events can lead to the production of anti-HLA memory B cells, but differ in terms of their inflammatory environment and the duration of allo-antigen exposure: pregnancy, transfusion or a previous transplantation. For the last group, the investigators want to distinguish two situations: kidney-transplanted patients that had an early transplantectomy due to thrombosis or that had an antibody-mediated rejection. Finally, patients can have anti-HLA antibodies without any sensitizing event identified. The investigators will first use an unbiased approach to test if anti-HLA memory B cells are heterogeneous. The investigators will perform single cell RNA sequencing of sorted anti-HLA B cells, identified with HLA tetramers, of five groups of patients based on their immunization histories. The investigators will further perform a phenotypic characterization of the tetramer+ anti-HLA B cells using spectral cytometry to study their nature and identify novel markers of memory subgroups.

ELIGIBILITY:
Inclusion Criteria:

* Adult kidney transplantation candidate at CHU de Bordeaux
* Sensitized against class I HLA
* Only on type of sensitizing event among : transfusion, pregnancy, previous transplantation, no senitizing event

Exclusion Criteria:

* Pediatric kidney transplantation candidate at CHU de Bordeaux
* Rituximab injection
* Ongoing treatment with immunosuppressive drugs
* Non-cutaneous carcinoma, chronic viral infection
* Acute infection
* Recent vaccination (<1 month)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2028-12-15 (Estimated)

PRIMARY OUTCOMES:
Memory B cell heterogeneity | At inclusion
  Memory B cell heterogeneity by single cell RNA sequencing

SECONDARY OUTCOMES:
Cytometry | At inclusion (Day 0), second visit (up to18 months) , third visit (up to 24 months)
  Memory B cell heterogeneity by flow cytometry

IPD SHARING:
Plan to Share IPD: No